CLINICAL TRIAL: NCT00967252
Title: An Observational Trial of Perioperative Atorvastatin on Inflammatory and Endothelial Function in Patients Undergoing Vascular Surgery (STAR-VaS 2)
Brief Title: Impact of Chronic Statin Use During Surgery on Inflammation and Infection Rates
Acronym: STAR-VaS2
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: David Neilipovitz MD FRCPC, The Ottawa Hospital
Other Study IDs: 2008526-01H
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Inflammation; Infection; Endothelial Function
Keywords: surgery; inflammation; infection; statins
MeSH Terms: conditions — Inflammation; Infections | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- atorvastatin 10 mg or equivalent dose: Patients already taking atorvastatin 10 mg or equivalent dose in another statin who is undergoing high risk surgery
  Interventions: Drug: Atorvastatin
- atorvastatin 20 mg or equivalent dose: Patients already taking atorvastatin 20 mg or equivalent dose in another statin who is undergoing high risk surgery
  Interventions: Drug: Atorvastatin
- atorvastatin 40 mg or equivalent dose: Patients already taking atorvastatin 40 mg or equivalent dose in another statin who is undergoing high risk surgery
  Interventions: Drug: Atorvastatin
- atorvastatin 80 mg or equivalent dose: Patients already taking atorvastatin 80 mg or equivalent dose in another statin who is undergoing high risk surgery
  Interventions: Drug: Atorvastatin
- non-statin group: Patients who are not taking or cannot take a statin drug who is undergoing high risk surgery
  Interventions: Other: Control

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10 mg daily or equivalent dose in another statin
  Other Names: lipitor
  Groups: atorvastatin 10 mg or equivalent dose
Drug: Atorvastatin — Atorvastatin 20 mg daily or equivalent dose in another statin
  Other Names: lipitor
  Groups: atorvastatin 20 mg or equivalent dose
Drug: Atorvastatin — Atorvastatin 40 mg daily or equivalent dose in another statin
  Other Names: lipitor
  Groups: atorvastatin 40 mg or equivalent dose
Drug: Atorvastatin — Atorvastatin 80 mg daily or equivalent dose in another statin
  Other Names: lipitor
  Groups: atorvastatin 80 mg or equivalent dose
Other: Control — No statin being taken
  Groups: non-statin group

SUMMARY:
Despite improvements in perioperative care, non-cardiac surgery remains associated with significant and costly complications. Analysis of perioperative deaths in the United Kingdom suggests that roughly 80% are directly attributable to infectious and cardiovascular complications. The best available evidence suggests that medical optimization is the preferred strategy to reduce cardiac risks but there has been no novel strategy to reduce nosocomial infection rates in over 20 years.

Emerging evidence in both the non-operative and operative setting suggest that statin drugs may prevent both infectious and cardiac events. The mechanism(s) of action are not entirely clear but appear to independent of lipid lowering effects and are often referred to as pleiotropic effects. Two key elements of the pleiotropic effects of statins appear to be their anti-inflammatory properties and improved endothelial vascular reactivity. The statin dose required to maximize these effects is unknown. A large observational trial suggests a contradictory dose effect with higher doses associated with reduced infectious complications and lower doses associated with fewer cardiac complications. Doctors therefore still have many unanswered questions about the use of statins in the perioperative setting. Should they be routinely started on all or only certain surgical patients? What dose of statin should be used? If a patient is already on a statin, should their dose be altered perioperatively? The latter question is particularly relevant in light of the marked increase in statin use. Recruitment logs for an ongoing trial demonstrate that over 70% of patients undergoing high-risk surgery were taking a statin but at markedly variable doses. This population presents an ideal opportunity to determine if there is a dose response relationship between statins and pleiotropic effects. We therefore propose an observational study that will determine anti-inflammatory and endothelial effects in high-risk surgical patients on varying doses of a perioperative statin drug.

Atorvastatin diminishes the rise in C-reactive protein (CRP), measured 48 hours after elective vascular surgery, in a dose dependent fashion.

Secondary Hypotheses:

Atorvastatin reduces endothelial dysfunction after elective vascular surgery, as measured by brachial artery ultrasound, in a dose dependent fashion.

DETAILED DESCRIPTION:
It is estimated that approximately 1.7 million surgical procedures are performed each year in Canada. Unfortunately, perioperative complications are not an uncommon occurrence and have substantial morbidity, mortality and costs associated with them. To date, the best strategies to reduce nosocomial infections are aseptic practices, timely prophylactic antibiotics and good surgical technique. Despite these strategies, it is estimated that at least 1 in 5 major vascular surgical patients will have some type of nosocomial infection within 30 days of their procedure. The direct and indirect mortality of infections in this population is difficult to estimate but nosocomial infections are estimated to contribute to at least 15% of the mortality in hospitalized patients.

The primary manner in which infections contribute to patient mortality is by progression to sepsis. Sepsis is the tenth leading cause of death in Canadians and worldwide is increasing in incidence and severity. The associated mortality of sepsis varies by population and infection source but is usually between 30-60%. Despite significant improvements in the management of sepsis in the last 5 years, there is still no generally effective preventive medication or strategy. Although cardiovascular complications, including myocardial infarction and heart failure, are less common at 15% of major vascular patients, they have a staggering mortality of around 30-50%. Clearly, strategies or therapies to reduce these complications could have profound benefits. The questions are therefore whether statin drugs reduce sepsis, cardiovascular complications, or both and, if they do, how might they do so.

Understanding of the pathophysiology of sepsis and acute coronary syndromes in the non-operative setting has led to tremendous advancements in the management. In sepsis, an excessive, inappropriate and misguided response in the host defense response is likely responsible. Massive cytokine release exacerbates endothelium dysfunction that then impacts coagulation, thrombolysis, inflammation, tissue repair and tissue growth. If not corrected, the endothelial cells either die directly or through the triggering of apoptosis. This then leads to multiorgan dysfunction and ultimately death. How sepsis ultimately impairs and damages endothelial cell function is likely multifactoral. Impairment of endothelial nitric oxide synthetase occurs that causes impaired perfusion and inappropriate microvasculature coagulation.

In a strikingly similar manner to sepsis, key elements to acute coronary syndromes again appear to be inflammation and endothelial dysfunction. Rupture of coronary plaques and thrombosis are central. Although perioperative myocardial events are traditionally said to be supply-demand problems, this theory is in dispute and evidence suggests that perioperative problems are very similar to non-operative events. Elevated levels of various inflammatory markers, particularly C-Reactive Protein, are associated with adverse cardiovascular events. Similarly, the vascular endothelium is responsible for regulating vasomotor tone, thrombosis, platelet and leukocyte interactions. Dysfunction of the endothelium is also believed to be a central component of the development of coronary complications. Although endothelial dysfunction has not been extensively investigated in the perioperative setting, pathophysiologic similarities make it probable that perioperative endothelial dysfunction contributes to the occurrence of perioperative myocardial events. Thus, strategies designed to control perioperative inflammation, as well as to improve endothelial function and stabilize coronary plaque have the potential to reduce both perioperative coronary and infectious events.

Although studies in both animals and humans strongly suggest that statins may both prevent and treat sepsis, no prospective randomized trials in humans have been conducted to demonstrate these effects. Although some statins have been demonstrated to directly attenuate replication and infectivity of microorganisms, the evidence primarily suggests that if statins are indeed protective it will likely be due to their anti-inflammatory and favorable endothelial effects. Improvement of endothelial function by statins has been suggested to prevent cardiac events by stabilizing coronary plaques and may even contribute to plaque regression. Statins restore endothelial production of endogenous nitric oxide synthetase thus improving organ perfusion and microvasculature thrombosis that is impaired in the setting of sepsis.

The goals of the proposed trial, STAR VaS II are therefore twofold: First, it will help determine if statin blunts the adverse perioperative changes in inflammation and endothelial function in a dose-dependent fashion. Second, it will determine if patients chronically on lower than maximal statin dose should have their dose increased in the perioperative period. We will evaluate the influence of varying doses of statins on perioperative inflammation, as assessed by C-reactive protein, and endothelial function as assessed by brachial artery ultrasound. If atorvastatin, chronically administered before surgery, improves inflammatory changes or endothelial function in a dose dependent fashion, then it is plausible that patients chronically on lower statin doses should have their dose increased in the perioperative period. If however patients on lower doses experienced similar benefit, as those on higher doses, then conceivably the recommended perioperative dose could be lower thereby theoretically further improving the risk-benefit ratio for a statin drug. All patients will be assessed for infections as defined by the CDC.

ELIGIBILITY:
Inclusion Criteria:

* over 45 years of age
* able to have a baseline brachial ultrasound test before their day of surgery
* elective high-risk surgery defined by use of the POISE criteria

Exclusion Criteria:

* lack of informed consent
* pregnant
* contraindication to the brachial artery ultrasound test protocol (i.e. contraindication to 0.4 mg sublingual nitroglycerin)
* enrolled in another conflicting study
* previously enrolled in STAR-VaS or STAR-VaS2

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective non-cardiac high-risk surgery as defined by the POISE criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
C-reactive protein levels | 48 hours postoperatively

SECONDARY OUTCOMES:
brachial artery reactivity (assessed by ultrasound) | preoperative compared to 24 hours postoperatively
Infection | 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: David T Neilipovitz, MD, Principal Investigator — The Ottawa Hospital; Greg L Bryson, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada